CLINICAL TRIAL: NCT00005222
Title: Decline in Cardiovascular Mortality: Framingham 1950-1984
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1101; R01HL040423 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases

SUMMARY:
To investigate possible mechanisms responsible for the decline in cardiovascular disease mortality among the Framingham Heart Study population and to evaluate the health status of survivors in terms of subsequent illness and functional limitations.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease mortality has declined more than 30 percent in the last thirty years. Almost two-thirds of this decline occurred between 1970 and 1980. Despite this decreased mortality, cardiovascular disease is still the leading cause of death. It is also the disease category associated with the most rapidly rising health care costs. Secular trends in lifestyle, self-care, improved access to medical care, and improvements in diagnostic and curative medicine have all been implicated. An understanding of the mechanisms contributing to this decline is necessary in order to develop a scientific basis for palliative and preventive care. Also, the dramatic decline in cardiovascular disease mortality has raised the issue of the quality of life among the survivors. The question is raised whether more people are surviving but with worsening health in terms of increased incidence and prevalence of disease as well as increased levels of functional limitation.

DESIGN NARRATIVE:

Five hypotheses were tested to address the issue of secular trends in lifestyle, self-care and medical care which may have influenced cardiovascular disease mortality. These were: differences in risk factor levels among similarly-aged birth cohorts influenced mortality by lessening the severity of disease or by improving recuperative capacity; mortality among the later birth cohorts declined due to less comorbid disease at the time of the disease event; long-term case fatality declined because the progression of disease was slower as evidenced by a reduction in disease recurrence; medical intervention reduced mortality by eliminating lethal sequelae in the later birth cohorts; decreased mortality resulted from medical innovations in diagnosis and therapy. Three hypotheses were tested to address the issue of worsening health among the survivors in the later birth cohorts. These were: although more individuals in the later birth cohorts survived 13 years of follow-up than did members of similarly-aged birth cohorts in earlier periods, they had higher rates of morbidity and were hospitalized more often; survivors in the later cohorts exhibited more disability in functional limitations; more survivors in the later cohorts were institutionalized in chronic care hospitals or skilled nursing facilities. Data on risk factors, co-morbidity, and recurrent cardiovascular disease in the three birth cohorts were already computerized. Data on medical interventions, improvement in case management, and the use of various technological innovations were abstracted from medical records and linked with the data on disease events. Data on functional limitations were available both by type and extent of disability from the Disability Analysis of Health Data, a study supported by the Social Security Administration. This data file was merged with the file for disease events to determine if general differences in functional health existed among the three birth cohorts at intake, and if between-cohort differences existed among survivors.

The study was renewed as a Shannon Award in Fiscal 1991.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1996-03 (Actual)